CLINICAL TRIAL: NCT00405990
Title: Optimizing the Impact of Prevention of Mother to Child Transmission of HIV in South Africa: the Forgotten Half of the Equation.
Brief Title: Male Partner Involvement in the Prevention of MTCT of HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Cape Town (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: cro625
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections
Keywords: HIV; MTCT; heterosexual behaviour; sexual risk behaviour; couple counselling; Voluntary counselling and testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Voluntary counselling and HIV testing in ANC for PMTCT — VCT for 30 minutes in ANC
  Other Names: ANC VCT; VCT for PMTCT
Behavioral: VCT — HIV VCT for PMTCT
  Other Names: VCT for PMTCT

SUMMARY:
The study aims to invite male sexual partners to attend antenatal clinic with their pregnant partners to either acquire pregnancy information or undergo voluntary counselling and testing for HIV. To see if male sexual partner involvement will decrease sexual risk behaviour.

DETAILED DESCRIPTION:
We will enrol 1000 pregnant women; recruited from antenatal clinic at Khayelitsha Midwive and Obstetric Unit (MOU). Community sensitization activities will be implemented in the catchment community to encourage male partner participation.

At the booking visit all women will be offered antenatal care, HIV group education and VCT as usual. Thereafter women will be recruited to enrol into the study, after signing the consent form half of the cohort members will be randomly assigned to partner VCT (Group A) and half to partner pregnancy information (Group B). Men in group B will be offered VCT at the second interview late in pregnancy. However, VCT will be provided if requested by study participants at any stage of the study or if the female partner is HIV positive. Women in group A will be given a written invitation to hand to their partners to encourage them to invite their partners to come to the antenatal clinic for VCT. In group B, women will be given a written invitation to give to their partners to encourage their partners to attend a pregnancy information session at the antenatal clinic.

VCT will be offered again close to delivery for all women and men who were previously uninfected or of unknown status. For those found to be HIV-infected at a prior visit, CD4 and CD8 T-cell counts, viral load, and full blood count tests will be conducted. Both women and men will be referred to the Antiretroviral clinic where ARV will be offered if appropriate and formula feeding (or exclusive breastfeeding) will be recommended. Reasons for declining VCT and data on sexual behaviour and violence will be sought at each visit.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for participation, a woman must be less than 30 weeks pregnant at enrolment.

Exclusion Criteria:

* Women who are more than 30 weeks pregnant will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Percentage of partners agreeing to attend VCT. | 12 weeks

SECONDARY OUTCOMES:
Percentage of partners and pregnant women abstaining, faithful to one partner and using condoms consistently. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boshishi K Mohlala, MBCHB FCOG MSC, Principal Investigator — Imperial College London
Locations (1):
- Khayelitsha Midwive and Obstetric Unit Site B, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Mohlala BK, Boily MC, Gregson S. The forgotten half of the equation: randomized controlled trial of a male invitation to attend couple voluntary counselling and testing. AIDS. 2011 Jul 31;25(12):1535-41. doi: 10.1097/QAD.0b013e328348fb85. PMID 21610487